CLINICAL TRIAL: NCT04350658
Title: Feasibility and Safety of TAVI Without Predilatation: an Observational All Comers Study
Brief Title: TAVR Without Predilatation
Acronym: TAVIWOP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0204
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Aortic Stenosis
Keywords: TAVR; Balloon prediltation; success of crossing the valve; direct implanation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVR: all comers study including all transfemoral or transcarotid TAVR procédures. direct implantation is the default strategy usually used in our enter as in may centers
  Interventions: Procedure: Transcatheter aortic valve implantation required for symptomatic aortic stenosis

INTERVENTIONS:
Procedure: Transcatheter aortic valve implantation required for symptomatic aortic stenosis — The procedure is performed via transfemoral or transcarotid access; Patients were confirmed to be eligible for TAVR by a multidisciplinary heart team including at least an interventional cardiologist, a cardiothoracic surgeon and an anesthetist. All TAVR implantation procedures were performed with the Edwards SAPIEN 3 THV or the MEDTRONIC CoreValve EVOLUT . For all patients, both vascular access and aortic valve were evaluated before the procedure by multislice computerized tomographic angiography (MSCT) of the entire aorta using vascular windows settings. The prosthesis and the vascular access were left to the discretion of the operating team. Transfemoral access was the first choice when possible. All TAVR procedures were performed in the same hybrid room (in Montpellier University Hospital), Most TAVR were performed under sedation or general anesthesia using mild low profile 14-16 French delivery systems and using percutaneous or surgical vascular access.

SUMMARY:
The procedure is performed via transfemoral or transcaprotid access; Patients were confirmed to be eligible for TAVR by a multidisciplinary heart team including at least an interventional cardiologist, a cardiothoracic surgeon and an anesthetist. All TAVR implantation procedures were performed with the Edwards SAPIEN 3 THV or the MEDTRONIC CoreValve EVOLUT . For all patients, both vascular access and aortic valve were evaluated before the procedure by multislice computerized tomographic angiography (MSCT) of the entire aorta using vascular windows settings. The prosthesis and the vascular access were left to the discretion of the operating team. Transfemoral access was the first choice when possible. All TAVR procedures were performed in the same hybrid room (in Montpellier University Hospital), Most TAVR were performed under sedation or general anesthesia using mild low profile 14-16 French delivery systems and using percutaneous or surgical vascular access.

ELIGIBILITY:
Inclusion criteria:

- patients undergoing TAVR via transfemoral or rascoarotid access

Exclusion criteria:

- others access (subclavian, apical, transaortic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all comers patients undergoing TAVR using transfemoral or transcaorotid approaches
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
success of the direct implantation | 1 day
  success of the direct implantation defined as failure of crossing with the THV after 3 attemps and absence of complication related to the direct crossing

SECONDARY OUTCOMES:
Indidence of post dilatation | 1 day
  Indidence of post dilatation
Underexpansion of the Edwards SAPIEN 3 THV | 1 day
  Underexpansion of the Edwards SAPIEN 3 THV
risks factors of failure of crossing | 1 day
  risks factors of failure of crossing : femoral vs carotid access, type of THV , vascular tortuosities, biscuipid valve, calcification, tight stenosis, horizontal aorta, small annulus

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC